CLINICAL TRIAL: NCT03180008
Title: Comparative Effectiveness of Customary Fit and Strong! vs. Fit and Strong Plus!
Brief Title: Fit and Strong! Plus Comparative Effectiveness Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Susan Hughes, Professor, Director, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0277; 1R01AG039374 (NIH)
Record Dates: First submitted 2017-05-30; First posted 2017-06-07 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis; Overweight and Obesity
MeSH Terms: conditions — Osteoarthritis; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fit and Strong! (Active Comparator): Fit & Strong! is evidence-based group exercise and self-management program. Classes meet for 90 minutes and include 60 minutes of physical activity (stretching/flexibility, low impact aerobics, and lower-extremity strength training) and 30 minutes of health education that follows a structured, scripted curriculum that centers on physical activity and osteoarthritis and incorporates self-efficacy, social support, and self-regulation. Classes are held 3 days per week for 8 weeks (24 sessions total).
  Interventions: Behavioral: Fit and Strong!
- Fit and Strong! Plus (Experimental): Fit & Strong! Plus differs from Fit & Strong! only in that the 30 minutes of health education, while retaining the core physical activity and osteoarthritis components, has weight and diet-related topics added to the curriculum.
  Interventions: Behavioral: Fit and Strong! Plus

INTERVENTIONS:
Behavioral: Fit and Strong! — Fit and Strong! is a group exercise and self-management program that meets for 90 minutes, 3 days per week, for 8 weeks. Each 90 minute session consists of 60 minutes of multi-component physical activity (stretching/flexibility exercises, low-impact aerobics, and strength/resistance exercise) and 30 minutes of health education delivered from a structured curriculum. The health education topics build self-efficacy for managing arthritis through physical activity.
  Arms: Fit and Strong!
Behavioral: Fit and Strong! Plus — The intervention consists of the traditional Fit and Strong! intervention (see previous description), but the health education component has been revised to focus on diet and weight management in addition to physical activity and arthritis.
  Arms: Fit and Strong! Plus

SUMMARY:
This randomized controlled trial is comparing outcomes of customary Fit and Strong!, to Fit and Strong! Plus, an enhanced version of the program that incorporates weight management. We hypothesize that Fit and Strong! Plus participants will show improved diet behaviors at 2, 6, 12, and 18 months that will be accompanied by a significant 5% weight loss at 6 months and maintained to 18 months, compared to participants in customary Fit and Strong!.

ELIGIBILITY:
Inclusion Criteria:

* Presence of symptoms of lower extremity osteoarthritis
* Age 60 or older
* Not currently participating in a regular physical activity program
* BMI 25-50
* Able to attend Fit and Strong! classes

Exclusion Criteria:

* Score of 3 or greater on Mental Status Questionnaire
* Recent hip or knee surgery
* Recent steroid injection into hip or knee
* Diagnosis of rheumatoid arthritis
* Uncontrolled diabetes
* Unspecified health conditions that may interfere with exercise

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hughes, DSW, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith-Ray RL, Fitzgibbon ML, Tussing-Humphreys L, Schiffer L, Shah A, Huber GM, Braunschweig C, Campbell RT, Hughes SL. Fit and Strong! Plus: design of a comparative effectiveness evaluation of a weight management program for older adults with osteoarthritis. Contemp Clin Trials. 2014 Mar;37(2):178-88. doi: 10.1016/j.cct.2013.11.014. Epub 2013 Dec 5. PMID 24316240
- [Background] Mears M, Tussing-Humphreys L, Cerwinske L, Tangney C, Hughes SL, Fitzgibbons M, Gomez-Perez S. Associations between Alternate Healthy Eating Index-2010, Body Composition, Osteoarthritis Severity, and Interleukin-6 in Older Overweight and Obese African American Females with Self-Reported Osteoarthritis. Nutrients. 2018 Dec 22;11(1):26. doi: 10.3390/nu11010026. PMID 30583501
- [Background] Fitzgibbon ML, Tussing-Humphreys L, Schiffer L, Smith-Ray R, Demott AD, Martinez M, Berbaum ML, Huber GM, Hughes SL. FIT & STRONG! PLUS: DESCRIPTIVE DEMOGRAPHIC AND RISK CHARACTERISTICS IN A COMPARATIVE EFFECTIVENESS TRIAL FOR OLDER AFRICAN-AMERICAN ADULTS WITH OSTEOARTHRITIS. J Aging Res Clin Pract. 2018;7(1):9-16. doi: 10.14283/jarcp.2018.3. PMID 30167430
- [Result] Hughes SL, Tussing-Humphreys L, Schiffer L, Smith-Ray R, Marquez DX, DeMott AD, Berbaum ML, Fitzgibbon ML. Fit & Strong! Plus Trial Outcomes for Obese Older Adults with Osteoarthritis. Gerontologist. 2020 Apr 2;60(3):558-570. doi: 10.1093/geront/gny146. PMID 30476065
- [Derived] Fitzgibbon ML, Tussing-Humphreys L, Schiffer L, Smith-Ray R, Marquez DX, DeMott AD, Berbaum ML, Hughes SL. Fit and Strong! Plus: Twelve and eighteen month follow-up results for a comparative effectiveness trial among overweight/obese older adults with osteoarthritis. Prev Med. 2020 Dec;141:106267. doi: 10.1016/j.ypmed.2020.106267. Epub 2020 Oct 3. PMID 33022324

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fit and Strong! | Fit and Strong! Plus
Started | 210 | 203
2-Month Follow-up | 192 | 191
6-Month Follow-up | 173 | 175
12-Month Follow-up | 169 | 156
Completed (18-Month Follow-up) | 182 | 174
Not Completed | 28 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fit and Strong! | Fit and Strong! Plus | Total
Number analyzed (Participants) | 210 | 203 | 413
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68 (6) | 68 (6) | 68 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 177 | 355
  Male | 32 | 26 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 202 | 195 | 397
  Unknown or Not Reported | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 193 | 187 | 380
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 210 | 203 | 413

OUTCOME MEASURES:

1. Primary Outcome: Dietary Intake
Description: The Healthy Eating Index 2010 (HEI-2010) measures diet quality based on the Dietary Guidelines for Americans. HEI-2010 total scores range from 0 to 100 points, with a higher score signifying superior diet quality.
Time Frame: 2, 6, 12, and 18 months
Population: The number analyzed at each time point varies due to loss to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Fit and Strong! | Fit and Strong! Plus
Number analyzed (Participants) | 210 | 203
score on a scale
  2-Month Follow-up: number analyzed (Participants) | 192 | 191
  2-Month Follow-up | 2.1 (0.7) | 4.7 (0.7)
  6-Month Follow-up: number analyzed (Participants) | 173 | 175
  6-Month Follow-up | 0.8 (0.7) | 2.0 (0.7)
  12-Month Follow-up: number analyzed (Participants) | 169 | 156
  12-Month Follow-up | 1.3 (0.7) | 0.6 (0.7)
  18-Month Follow-up: number analyzed (Participants) | 182 | 174
  18-Month Follow-up | 0.0 (0.7) | 1.0 (0.7)

2. Primary Outcome: Body Weight
Description: A change in body weight (kilograms) measured using a calibrated digital scale (Tanita).
Time Frame: 2, 6, 12, and 18 months
Population: The number analyzed at each time point varies due to loss to follow-up.
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Fit and Strong! | Fit and Strong! Plus
Number analyzed (Participants) | 210 | 203
Kilograms
  2-Month Follow-up: number analyzed (Participants) | 192 | 191
  2-Month Follow-up | -0.5 (0.2) | -2.0 (0.2)
  6-Month Follow-up: number analyzed (Participants) | 173 | 175
  6-Month Follow-up | -0.8 (0.3) | -2.0 (0.3)
  12-Month Follow-up: number analyzed (Participants) | 169 | 156
  12-Month Follow-up | -0.9 (0.3) | -1.7 (0.3)
  18-Month Follow-up: number analyzed (Participants) | 182 | 174
  18-Month Follow-up | -0.9 (0.3) | -1.3 (0.3)

3. Secondary Outcome: Physical Activity Engagement
Description: A change in Physical activity was assessed using the Physical Activity Scale for the Elderly (PASE). Scored on a scale of 0 - 400, a higher score indicates greater PA.
Time Frame: 2, 6, 12, and 18 months
Population: The number analyzed at each time point varies due to loss to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Fit and Strong! | Fit and Strong! Plus
Number analyzed (Participants) | 210 | 203
score on a scale
  2 months: number analyzed (Participants) | 192 | 191
  2 months | 14.1 (4.7) | 29.1 (4.8)
  6 months: number analyzed (Participants) | 173 | 175
  6 months | 15.4 (5.0) | 17.5 (5.0)
  12 months: number analyzed (Participants) | 169 | 156
  12 months | 7.0 (4.8) | 11.6 (4.9)
  18 months: number analyzed (Participants) | 182 | 174
  18 months | 5.2 (4.8) | 12.2 (4.9)

4. Secondary Outcome: Lower Extremity Pain
Description: A change in Osteoarthritis "lower extremity pain" symptoms were measured using the Western Ontario and McMaster Universities Arthritis Index (WOMAC). The WOMAC is a self-report instrument that has been well-validated and used widely with individuals with osteoarthritis. Pain (5 items) was rated on a Likert scale ranging from 0 (none) to four. Higher scores indicate more severe osteoarthritis symptoms, scores range from 0-20.
Time Frame: Baseline, 2, 6, 12, and 18 months
Population: The number analyzed at each time point varies due to loss to follow-up.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Fit and Strong! | Fit and Strong! Plus
Number analyzed (Participants) | 210 | 203
Score on a scale
  2-Month Follow: number analyzed (Participants) | 192 | 191
  2-Month Follow | -0.5 (0.2) | -1.4 (0.2)
  6-Month: number analyzed (Participants) | 173 | 175
  6-Month | -0.6 (0.3) | -1.5 (0.3)
  12-Month: number analyzed (Participants) | 169 | 156
  12-Month | -0.7 (0.3) | -0.9 (0.3)
  18-Month: number analyzed (Participants) | 182 | 174
  18-Month | -0.1 (0.3) | -0.9 (0.3)

5. Secondary Outcome: Lower Extremity Stiffness
Description: A change in Osteoarthritis "lower extremity stiffness" symptoms were measured using the Western Ontario and McMaster Universities Arthritis Index (WOMAC). The WOMAC is a self-report instrument that has been well-validated and used widely with individuals with osteoarthritis. Stiffness (2 items) was rated on a Likert scale ranging from 0 (none) to four. Higher scores indicate more severe osteoarthritis symptoms, scores range from 0 to 8.
Time Frame: Baseline, 2, 6, 12, and 18 months
Population: The number analyzed at each time point varies due to loss to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Fit and Strong! | Fit and Strong! Plus
Number analyzed (Participants) | 210 | 203
score on a scale
  2-Month: number analyzed (Participants) | 192 | 191
  2-Month | -0.3 (0.1) | -0.6 (0.1)
  6-Month: number analyzed (Participants) | 173 | 175
  6-Month | -0.5 (0.1) | -0.5 (0.1)
  12-Month: number analyzed (Participants) | 169 | 156
  12-Month | -0.6 (0.1) | -0.5 (0.1)
  18-Month: number analyzed (Participants) | 182 | 174
  18-Month | -0.6 (0.1) | -0.4 (0.1)

6. Secondary Outcome: Lower Extremity Physical Function
Description: A change in Osteoarthritis "lower extremity physical function" symptoms were measured using the Western Ontario and McMaster Universities Arthritis Index (WOMAC). The WOMAC is a self-report instrument that has been well-validated and used widely with individuals with osteoarthritis. Lower extremity physical function (17 items) was rated on a Likert scale ranging from 0 (none) to four. Higher scores indicate more severe osteoarthritis symptoms, scores range from 0 to 68.
Time Frame: Baseline, 2, 6, 12, and 18 months
Population: The number analyzed at each time point varies due to loss to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Fit and Strong! | Fit and Strong! Plus
Number analyzed (Participants) | 210 | 203
score on a scale
  2-Month: number analyzed (Participants) | 192 | 191
  2-Month | -1.9 (0.7) | -5.5 (0.8)
  6-Month: number analyzed (Participants) | 173 | 175
  6-Month | -1.7 (0.9) | -4.9 (0.9)
  12-Month: number analyzed (Participants) | 169 | 156
  12-Month | -2.0 (0.9) | -4.1 (0.9)
  18-Month: number analyzed (Participants) | 182 | 174
  18-Month | -2.6 (0.9) | -3.5 (0.9)

7. Secondary Outcome: Lower Extremity Muscle Strength
Description: A change in Lower Extremity Muscle Strength was measured by a Sit-Stand test that measures the number of full stands from a seated position a participant can complete in 30 s with arms folded across the chest. A higher score reflects better performance.
Time Frame: Baseline, 2, 6, 12, and 18 months
Population: The number analyzed at each time point varies due to loss to follow-up.
Measure: Mean (Standard Error); unit: number of chair stands
Arm/Group | Fit and Strong! | Fit and Strong! Plus
Number analyzed (Participants) | 210 | 203
number of chair stands
  2-Month: number analyzed (Participants) | 192 | 191
  2-Month | 1.3 (0.2) | 1.8 (0.2)
  6-Month: number analyzed (Participants) | 173 | 175
  6-Month | 1.1 (0.2) | 1.7 (0.2)
  12-Month: number analyzed (Participants) | 169 | 156
  12-Month | 1.0 (0.2) | 1.6 (0.2)
  18-Month: number analyzed (Participants) | 182 | 174
  18-Month | 0.7 (0.2) | 1.4 (0.2)

8. Secondary Outcome: Physical Endurance
Description: A change in Physical Endurance was measured by the 6-minute Distance Walk, which is a self-paced timed test of the total distance a person can walk in six minutes. A higher score reflects better performance.
Time Frame: Baseline, 2, 6, 12, and 18 months
Population: The number analyzed at each time point varies due to loss to follow-up.
Measure: Mean (Standard Error); unit: meters walked
Arm/Group | Fit and Strong! | Fit and Strong! Plus
Number analyzed (Participants) | 210 | 203
meters walked
  2-Month: number analyzed (Participants) | 192 | 191
  2-Month | 22.9 (4.4) | 50.5 (4.4)
  6-Month: number analyzed (Participants) | 173 | 175
  6-Month | 13.3 (5.2) | 29.3 (5.1)
  12-Month: number analyzed (Participants) | 169 | 156
  12-Month | 10.0 (5.3) | 23.2 (5.3)
  18-Month: number analyzed (Participants) | 182 | 174
  18-Month | -0.6 (5.8) | 12.8 (5.8)

ADVERSE EVENTS:
Time Frame: 18 months.
Arm/Group | Fit and Strong! | Fit and Strong! Plus
All-Cause Mortality (participants affected / at risk) | 3/210 | 4/203
Serious Adverse Events (participants affected / at risk) | 1/210 | 0/203
Other Adverse Events (participants affected / at risk) | 1/210 | 4/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fit and Strong! (N=210) | Fit and Strong! Plus (N=203)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Participant fell on ice, due to winter weather, outside of study site for follow-up visit. No serious or lasting injuries reported.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fit and Strong! (N=210) | Fit and Strong! Plus (N=203)
Feeling faint/lightheaded (General disorders) | 1 (1) | 1 (1) — Feeling faint/lightheaded while exercising, not resulting in injury or other problems.
Discomfort during exercise (General disorders) | 0 (0) | 3 (3) — Reports of feeling pain/discomfort during or resulting from exercise, without serious injury or other problems

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT03180008/Prot_SAP_000.pdf